CLINICAL TRIAL: NCT03907033
Title: Preemptive Local Analgesia With Liposomal Bupivacaine in Vaginal Hysterectomy: A Randomized Controlled Study
Brief Title: Liposomal Bupivacaine in Vaginal Hysterectomy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient funding to continue with study activities
Sponsor: Mayo Clinic (Other)
Collaborators: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Principal Investigator, Johnny Yi, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 15-008413
Record Dates: First submitted 2019-04-05; First posted 2019-04-08 (Actual); Results first posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-09

CONDITIONS: Vaginal Hysterectomy
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to receive either the bupivacaine HCl injection at the time of surgery or bupivacaine HCl plus liposomal bupivacaine.
Who Masked: Participant, Care Provider, Investigator
Masking Description: This will be a blinded study where investigators, patients, and care providers will be blinded to treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Bupivacaine (Active Comparator): Patients in the control group will receive 0.25% bupivacaine hydrochloride (bupivacaine HCl). 10cc will be injected bilaterally into each uterosacral ligament prior to the colpotomy incision. After entry into the posterior cul-de-sac, an additional 10cc of will be injected bilaterally into the deeper uterosacral ligaments.
  Interventions: Drug: Bupivacaine Hydrochloride
- Liposomal Bupivacaine (Experimental): Patients in the study group will receive a mixture of 0.5% bupivacaine HCl and liposomal bupivacaine in 1:1 ratio. 10cc of the mixture will be injected bilaterally into each uterosacral ligament prior to the colpotomy incision. After entry into the posterior cul-de-sac, an additional 10cc will be injected bilaterally into the deeper uterosacral ligaments
  Interventions: Drug: Liposomal bupivacaine; Drug: Bupivacaine Hydrochloride

INTERVENTIONS:
Drug: Liposomal bupivacaine — Liposomal bupivacaine is a novel formulation of local bupivacaine and allows prolonged release of the medication, thereby providing longer lasting effects. It is approved by the FDA and has been shown to provide excellent pain control after surgery.
  Other Names: Exparel
  Arms: Liposomal Bupivacaine
Drug: Bupivacaine Hydrochloride — We currently administer local plain bupivacaine during vaginal hysterectomy to decrease pain in the postoperative period. Bupivacaine is an anesthetic that works by blocking nerve conduction and producing a numbing effect.

SUMMARY:
The aim of this study is to compare the effects of preemptive analgesia using liposomal bupivacaine mixed with bupivacaine HCl, versus bupivacaine HCl alone for uterosacral ligament injection in patients undergoing vaginal hysterectomy. We hypothesize that the group receiving a combination of liposomal bupivacaine and bupivacaine HCl will report superior postoperative pain management. Enhancement in pain control should confer a decrease in opioid and other analgesic medication requirements, which may contribute to decreased nausea, vomiting, and higher overall patient satisfaction with pain control.

DETAILED DESCRIPTION:
Prior to surgery, patients are assigned by chance (like a coin toss) to receive either the bupivacaine HCl injection at the time of surgery or bupivacaine HCl plus liposomal bupivacaine. Patients and the Principal Investigator cannot choose the study group. Patients will have a 50% chance of being assigned to either group; however, regardless of which group they are assigned to, the medical record will show that they received liposomal bupivacaine. The injections will be given in the vaginal area when the patient is under anesthesia.

After surgery, patients will be asked to record their pain, medication use, pain scores and symptoms in a diary for each 12 hour interval up to 72 hours. Someone will also call twice a day during the 72 hours after surgery to ask about pain level and pain medication use.

Patients will also receive a phone call 7-10 days after the surgery to ask about their recovery and pain level.

ELIGIBILITY:
INCLUSION CRITERIA

1. Women 18-85 who will be having an outpatient vaginal hysterectomy with or without concurrent prolapse repair surgery at Mayo Clinic Hospital in Arizona

EXCLUSION CRITERIA

1. Known history of hepatic (liver) disease as evidenced by an AST or ALT that is greater than normal values
2. Known history of renal (kidney) disease as evidenced by a serum creatinine that is greater than normal values
3. Known history of prolonged QT (QTc greater than 500 m/s)
4. Opiate tolerance as noted by daily use of greater than 20 mg morphine daily oral equivalents per day for a minimum of 1 month prior to surgery
5. Allergy or contraindication to amide local anesthetics, celecoxib, ketorolac, NSAIDs, acetaminophen, gabapentin, sulfa drugs, or ondansetron
6. Allergy to both oxycodone and hydromorphone
7. Patients with acute gastrointestinal bleed that has occurred less than 6 months prior to study enrollment
8. Adults lacking the ability to consent

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2021-07-23 (Actual); Study Completion 2021-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Cornella, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Long JB, Eiland RJ, Hentz JG, Mergens PA, Magtibay PM, Kho RM, Magrina JF, Cornella JL. Randomized trial of preemptive local analgesia in vaginal surgery. Int Urogynecol J Pelvic Floor Dysfunct. 2009 Jan;20(1):5-10. doi: 10.1007/s00192-008-0716-6. Epub 2008 Oct 2. PMID 18830553
- [Background] Ilfeld BM, Viscusi ER, Hadzic A, Minkowitz HS, Morren MD, Lookabaugh J, Joshi GP. Safety and Side Effect Profile of Liposome Bupivacaine (Exparel) in Peripheral Nerve Blocks. Reg Anesth Pain Med. 2015 Sep-Oct;40(5):572-82. doi: 10.1097/AAP.0000000000000283. PMID 26204387
- [Background] Bergese SD, Ramamoorthy S, Patou G, Bramlett K, Gorfine SR, Candiotti KA. Efficacy profile of liposome bupivacaine, a novel formulation of bupivacaine for postsurgical analgesia. J Pain Res. 2012;5:107-16. doi: 10.2147/JPR.S30861. Epub 2012 May 1. PMID 22570563
- [Background] Hutchins J, Delaney D, Vogel RI, Ghebre RG, Downs LS Jr, Carson L, Mullany S, Teoh D, Geller MA. Ultrasound guided subcostal transversus abdominis plane (TAP) infiltration with liposomal bupivacaine for patients undergoing robotic assisted hysterectomy: A prospective randomized controlled study. Gynecol Oncol. 2015 Sep;138(3):609-13. doi: 10.1016/j.ygyno.2015.06.008. Epub 2015 Jun 6. PMID 26056753
- [Background] Mont MA, Beaver WB, Dysart SH, Barrington JW, Del Gaizo DJ. Local Infiltration Analgesia With Liposomal Bupivacaine Improves Pain Scores and Reduces Opioid Use After Total Knee Arthroplasty: Results of a Randomized Controlled Trial. J Arthroplasty. 2018 Jan;33(1):90-96. doi: 10.1016/j.arth.2017.07.024. Epub 2017 Jul 25. PMID 28802777
- [Background] Kalogera E, Bakkum-Gamez JN, Jankowski CJ, Trabuco E, Lovely JK, Dhanorker S, Grubbs PL, Weaver AL, Haas LR, Borah BJ, Bursiek AA, Walsh MT, Cliby WA, Dowdy SC. Enhanced recovery in gynecologic surgery. Obstet Gynecol. 2013 Aug;122(2 Pt 1):319-328. doi: 10.1097/AOG.0b013e31829aa780. PMID 23969801
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Bupivacaine | Liposomal Bupivacaine
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Bupivacaine | Liposomal Bupivacaine | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (10.96) | 60.4 (12.56) | 57.8 (11.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Total Post-surgical Opioid Medication Use
Description: Participants post-surgical analgesic medication use of IV hydrocodone and oxycodone measured in morphine equivalents (ME)
Time Frame: First 72 hours following surgery completion
Measure: Median (Full Range); unit: Morphine Equivalents (ME)
Arm/Group | Standard Bupivacaine | Liposomal Bupivacaine
Number analyzed (Participants) | 14 | 14
Morphine Equivalents (ME)
  Hydrocodone | 0 [0.0 to 0.0] | 0 [0.0 to 0.0]
  Oxycodone | 30.0 [0.0 to 82.5] | 30.0 [0.0 to 135.0]
Statistical Analysis 1: Comparison: Standard Bupivacaine vs Liposomal Bupivacaine; Standard Bupivacaine study arm compared to Liposomal Bupivacaine study arm for Hydrocodone use; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Standard Bupivacaine vs Liposomal Bupivacaine; Standard Bupivacaine study arm compared to Liposomal Bupivacaine study arm for Oxycodone use; Test type: Superiority; p = 0.010, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Total Post-surgical Analgesic Medication Use
Description: Participants post-surgical analgesic medication use of Ibuprofen and acetaminophen measured in milligrams (mg)
Time Frame: First 72 hours following surgery completion
Measure: Median (Full Range); unit: mg
Arm/Group | Standard Bupivacaine | Liposomal Bupivacaine
Number analyzed (Participants) | 14 | 14
mg
  Ibuprofen | 5400.0 [3000.0 to 13200.0] | 4800.0 [0.0 to 13200.00]
  Tylenol | 6500.0 [0.0 to 13000.0] | 6500.0 [500.0 to 13000.0]
Statistical Analysis 1: Comparison: Standard Bupivacaine vs Liposomal Bupivacaine; Standard Bupivacaine study arm compared to Liposomal Bupivacaine study arm for Ibuprofen use; Test type: Superiority; p = 0.248, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Standard Bupivacaine vs Liposomal Bupivacaine; Standard Bupivacaine study arm compared to Liposomal Bupivacaine study arm for Tylenol use; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Mean PACU Visual Analog Scale (VAS) (0-10) Pain Score
Description: Scale Ranges from 0 (no pain) to 10 (extreme pain)
Time Frame: Assessed while patient in PACU for recovery post-surgery per standard procedure
Population: Data not collected or analyzed
Arm/Group | Standard Bupivacaine | Liposomal Bupivacaine
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: VAS Pain Score at 24, 48, and 72 Hours Post-surgery Completion
Description: Scale Ranges from 0 (no pain) to 10 (extreme pain)
Time Frame: 24, 48, and 72 hours post-surgery completion
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Standard Bupivacaine | Liposomal Bupivacaine
Number analyzed (Participants) | 14 | 14
score on a scale
  24 hours post-surgery | 3.1 [1.0 to 7.5] | 3.5 [0.0 to 7.5]
  48 hours post-surgery | 2.5 [1.0 to 5.8] | 3.6 [0.0 to 9.0]
  72 hours post-surgery | 1.6 [0.3 to 4.5] | 2.4 [0.0 to 7.5]
Statistical Analysis 1: Comparison: Standard Bupivacaine vs Liposomal Bupivacaine; Standard Bupivacaine study arm compared to Liposomal Bupivacaine study arm 24 hours post-surgery; Test type: Superiority; p = 0.846, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Standard Bupivacaine vs Liposomal Bupivacaine; Standard Bupivacaine study arm compared to Liposomal Bupivacaine study arm 48 hours post-surgery; Test type: Superiority; p = 0.490, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Standard Bupivacaine vs Liposomal Bupivacaine; Standard Bupivacaine study arm compared to Liposomal Bupivacaine study arm 72 hours post-surgery; Test type: Superiority; p = 0.564, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Nausea at 24, 48, and 72 Hours Post-surgery Completion
Description: Number of times patient reported feeling nauseous
Time Frame: 24, 48, and 72 hours post-surgery
Measure: Median (Full Range); unit: events
Arm/Group | Standard Bupivacaine | Liposomal Bupivacaine
Number analyzed (Participants) | 14 | 14
events
  24 hours post-surgery | 0.0 [0.0 to 3.0] | 0.0 [0.0 to 22.0]
  48 hours post-surgery | 0.0 [0.0 to 6.0] | 0.0 [0.0 to 20.0]
  72 hours post-surgery | 0.0 [0.0 to 3.0] | 0.0 [0.0 to 14.0]
Statistical Analysis 1: Comparison: Standard Bupivacaine vs Liposomal Bupivacaine; Standard Bupivacaine study arm compared to Liposomal Bupivacaine arm at 24 hours post-surgery; Test type: Superiority; p = 0.264, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Standard Bupivacaine vs Liposomal Bupivacaine; Standard Bupivacaine study arm compared to Liposomal Bupivacaine arm at 48 hours post-surgery; Test type: Superiority; p = 0.970, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Standard Bupivacaine vs Liposomal Bupivacaine; Standard Bupivacaine study arm compared to Liposomal Bupivacaine arm at 72 hours post-surgery; Test type: Superiority; p = 0.536, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Emesis at 24, 48, and 72 Hours Post-surgery Completion
Description: Number of times the patient vomited
Time Frame: 24, 48, and 72 hours post-surgery
Measure: Median (Full Range); unit: events
Arm/Group | Standard Bupivacaine | Liposomal Bupivacaine
Number analyzed (Participants) | 14 | 14
events
  24 hours post-surgery | 0.0 [0.0 to 1.0] | 0.0 [0.0 to 2.0]
  48 hours post-surgery | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 1.0]
  72 hours post-surgery | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 11.0]
Statistical Analysis 1: Comparison: Standard Bupivacaine vs Liposomal Bupivacaine; Standard Bupivacaine study arm compared to Liposomal Bupivacaine study arm at 24 hours post-surgery; Test type: Superiority; p = 0.957, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Standard Bupivacaine vs Liposomal Bupivacaine; Standard Bupivacaine study arm compared to Liposomal Bupivacaine study arm at 48 hours post-surgery; Test type: Superiority; p = 0.353, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Standard Bupivacaine vs Liposomal Bupivacaine; Standard Bupivacaine study arm compared to Liposomal Bupivacaine study arm at 72 hours post-surgery; Test type: Superiority; p = 0.165, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Urinary Retention
Description: Number of patients who had post-void residual (PVR) >150cc's at voiding trial prior to discharge
Time Frame: At voiding trial prior to discharge from hospital, approximately 72 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Bupivacaine | Liposomal Bupivacaine
Number analyzed (Participants) | 14 | 14
Participants | 1 | 1

8. Secondary Outcome: Patient Satisfaction With Pain Management at 72 Hours and 7-10 Days Post Surgery
Description: Assessed on 0-10 scale (0 being worst level of satisfaction, 10 being best level)
Time Frame: 72 hours and 7-10 days post surgery
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Standard Bupivacaine | Liposomal Bupivacaine
Number analyzed (Participants) | 14 | 14
score on a scale
  72 hours post-surgery | 10.0 [5.0 to 10.0] | 9.5 [1.0 to 10.0]
  7-10 days post-surgery | 10.00 [7.0 to 10.0] | 9.0 [8.0 to 10.0]
Statistical Analysis 1: Comparison: Standard Bupivacaine vs Liposomal Bupivacaine; Standard Bupivacaine study arm compared to Liposomal Bupivacaine study arm at 72 hours post-surgery; Test type: Superiority; p = 0.802, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Standard Bupivacaine vs Liposomal Bupivacaine; Standard Bupivacaine study arm compared to Liposomal Bupivacaine study arm at 7-10 days post-surgery; Test type: Superiority; p = 0.656, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events were collected post operative on all participants, approximately 7 days.
Arm/Group | Standard Bupivacaine | Liposomal Bupivacaine
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 3/14 | 2/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Bupivacaine (N=14) | Liposomal Bupivacaine (N=14)
Urinary Retention (Renal and urinary disorders) | 1 | 1
Urinary Incontinence (Renal and urinary disorders) | 1 | 1
Protruding sutures (Surgical and medical procedures) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-27): https://cdn.clinicaltrials.gov/large-docs/33/NCT03907033/Prot_SAP_000.pdf